CLINICAL TRIAL: NCT07104448
Title: Impact of a Standardized Perioperative Care Protocol on Functional and Radiographic Outcomes Following Transforaminal Lumbar Interbody Fusion for Degenerative Spondylolisthesis: A Randomized Controlled Trial
Brief Title: Standardized Perioperative Care Protocol for Lumbar Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Principal Investigator, Baoli Li, Principal investigator, Hebei Medical University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE2017-011-1
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Degenerative Lumbar Spondylolisthesis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Standardized Perioperative Care Protocol (SPCP) Group (Experimental): Patients randomized to this group received a multi-modal, standardized protocol that included: comprehensive preoperative education and optimization; standardized intraoperative anesthesia and surgical techniques; and a structured postoperative rehabilitation program featuring multimodal analgesia and goal-directed early mobilization.
  Interventions: Behavioral: Standardized Perioperative Care Protocol
- Active Comparator: Conventional Care Group (Active Comparator): Patients randomized to this group received standard institutional care, which was not protocolized. This typically involved surgeon-preference-based perioperative management, variable timing for mobilization and catheter removal, and discharge based on the attending surgeon's general assessment.
  Interventions: Other: Conventional care

INTERVENTIONS:
Behavioral: Standardized Perioperative Care Protocol — A multi-component protocol involving preoperative patient education, nutritional screening, standardized anesthesia, goal-directed fluid therapy, multimodal opioid-sparing analgesia, and a structured physiotherapy-led mobilization schedule starting on postoperative day 1.
  Arms: Experimental: Standardized Perioperative Care Protocol (SPCP) Group
Other: Conventional care — Standard, non-protocolized institutional perioperative care, with management decisions based on the discretion of the attending surgeon and care team.
  Arms: Active Comparator: Conventional Care Group

SUMMARY:
This is a prospective, randomized controlled trial to evaluate whether a comprehensive, standardized perioperative care protocol (SPCP) improves functional recovery, radiographic outcomes, and quality of life compared to conventional care in patients undergoing transforaminal lumbar interbody fusion (TLIF) for degenerative lumbar spondylolisthesis. The study aims to demonstrate that a protocol-driven approach can lead to better patient outcomes and increased healthcare efficiency.

DETAILED DESCRIPTION:
Transforaminal lumbar interbody fusion (TLIF) is a common surgical treatment for degenerative lumbar spondylolisthesis, but patient outcomes can be variable due to inconsistencies in perioperative management. Enhanced Recovery After Surgery (ERAS) principles have shown promise, but their comprehensive application in spine surgery requires further validation. This study hypothesizes that a multifaceted Standardized Perioperative Care Protocol (SPCP), which integrates preoperative optimization (education, nutrition), standardized intraoperative techniques, and a structured, goal-directed postoperative rehabilitation plan, will result in superior outcomes compared to conventional, non-protocolized care. A total of 382 patients were randomized to either the SPCP or conventional care group. The study will assess outcomes at multiple time points up to 2 years post-surgery to determine the long-term efficacy of the protocol in improving functional recovery, spinal fusion, quality of life, and reducing complications.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, single-level (L3-L4, L4-L5, or L5-S1) degenerative spondylolisthesis (Meyerding Grade I or II).
* Failure of at least 6 months of conservative therapy.
* Age between 40 and 75 years.
* Suitable for and scheduled to undergo transforaminal lumbar interbody fusion (TLIF) surgery.
* Provided written informed consent.

Exclusion Criteria:

* High-grade spondylolisthesis (Grade > II).
* History of previous lumbar surgery.
* Presence of active spinal infection, tumor, or trauma.
* Severe osteoporosis (T-score < -3.0).
* Significant medical comorbidities precluding major surgery (ASA physical status > III).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) Score | Baseline, 2 years
  The change in the ODI score from baseline to 2 years post-surgery. The ODI (version 2.1a) is a patient-reported outcome measure that assesses disability due to low back pain. Scores range from 0 to 100, with lower scores indicating less disability.

SECONDARY OUTCOMES:
Change in Japanese Orthopaedic Association (JOA) Score | Baseline, 3 months, 6 months, 1 year, 2 years
  Change from baseline in the JOA score, which evaluates clinical symptoms, function, and activities of daily living for patients with lumbar disease. Scores range from 0-29, with higher scores indicating better function.
Change in Visual Analog Scale (VAS) for Back and Leg Pain | Baseline, 3 months, 6 months, 1 year, 2 years
  Change from baseline in patient-reported back and leg pain, measured on a 0-10 scale, where 0 represents no pain and 10 represents the worst imaginable pain.
Change in Short Form-36 (SF-36) Quality of Life Scores | Baseline, 3 months, 6 months, 1 year, 2 years
  Change from baseline in the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores of the SF-36 survey, which measures health-related quality of life.
Radiographic Fusion Rate | 1 year, 2 years
  The proportion of patients achieving solid fusion (Bridwell classification Grade I or II) at the index surgical level, as assessed by standing lateral X-rays.
Change in Segmental Lordosis | Baseline, 1 year, 2 years
  Change from baseline in the segmental lordosis angle at the index surgical level, measured on standing lateral X-rays.
Change in Posterior Disc Height | Baseline, 1 year, 2 years
  Change from baseline in the posterior disc height at the index surgical level, measured on standing lateral X-rays.
Length of Hospital Stay (LOS) | During hospital stay, up to approximately 14 days post-surgery
  The total number of days from admission to discharge for the index surgical procedure.
Incidence of Postoperative Complications | Up to 90 days post-surgery
  The number and proportion of patients experiencing any adverse events within 90 days of surgery, including but not limited to surgical site infection, dural tear, DVT, ileus, and urinary retention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Zhao Y, Wu J, Zhang Z, Wang Y, Li B. Impact of a standardized perioperative care protocol on functional and radiographic outcomes following transforaminal lumbar interbody fusion for degenerative spondylolisthesis: a 2-year randomized controlled trial. Front Surg. 2025 Dec 18;12:1679851. doi: 10.3389/fsurg.2025.1679851. eCollection 2025. PMID 41488876